CLINICAL TRIAL: NCT02365311
Title: Echocardiographic Evaluation of the Change on Pulmonary Blood Flow and Cardiac Function During One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 4-2014-0486
Record Dates: First submitted 2015-02-02; First posted 2015-02-18 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Video-assisted Thoracic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one lung group (Experimental)
  Interventions: Procedure: transesophageal echocardiography(TEE)

INTERVENTIONS:
Procedure: transesophageal echocardiography(TEE) — Transesophageal echocardiography examination will be performed TLV in supine and lateral position, 10, 20 and 30 min during OLV in left lateral decubitus position. By using the transesophageal echocardiography, we will evaluate the changes of pulmonary blood flow and cardiac function.

SUMMARY:
The investigators used transesophageal echocardiography (TEE) to assess the change of pulmonary blood flow and bi-ventricular function during lung isolation. The investigators hypothesized that changes in pulmonary venous flow with lung isolation may be related the shunt fraction and oxygenation during one lung ventilation (OLV). The investigators also observed the cardiac function during two lung ventilation (TLV) and OLV in supine and lateral position by TEE.

ELIGIBILITY:
Inclusion Criteria:

* Above 20 years of age.
* American Society of Anesthesiologists (ASA) Physical Status I and II
* Thoracic surgical procedure (video-assisted)

Exclusion Criteria:

* severe functional liver or kidney disease
* cardiac disease
* arrhythmia
* exceed BMI > 30 kg/ m2
* COPD
* pathologic esophageal lesion (esophageal stricture or varix )
* pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The change of pulmonary blood flow | two-lung ventilation in the supine (T1) and lateral position (T2) and 10 (T3), 20 (T4), and 30 min (T5) during OLV in the left lateral decubitus position.
  Pulmonary blood flow = PVA(cross sectional area of LUPV) x VTI(velocity time integral) x HR , Fractional area change = [(LVAd-LVAs)/LVAd] × 100 Ejection fraction = [(LVEDV(LV end-diastolic volume) -LVESV(LV end-systolic volume)/LVEDV] × 100

SECONDARY OUTCOMES:
The changes of respiratory parameters | two-lung ventilation in the supine (T1) and lateral position (T2) and 10 (T3), 20 (T4), and 30 min (T5) during OLV in the left lateral decubitus position.
  shunt fraction Qs/Qt = (CcO2- CaO2)/(CcO2- CvO2) CcO2 = Hgb x 1.34 x ScO2 + PcO2 x 0.003, lung compliance : Compliance= Vt / Pplat, physiologic dead space : Vd/Vt = 1.14 x (PaCO2 - PETCO2)/PaCO2- 0.005
The change of cardiac function | two-lung ventilation in the supine (T1) and lateral position (T2) and 10 (T3), 20 (T4), and 30 min (T5) during OLV in the left lateral decubitus position.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea